CLINICAL TRIAL: NCT04364932
Title: Antenatal and Intrapartum Risk Factors Associated With Neonatal Hypoxic Ischemic Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa Rady Ali, Resident doctor, Assiut University
Other Study IDs: HIE risk factors
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Neonatal Hypoxic Ischemic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perinatal asphyxia is a major cause of hypoxic Ischemic encephalopathy (HIE), perinatal death and long term neurodisability. This can be devastating for the individual and their family; the healthcare and litigation costs notwithstanding. In recent years have attempted to quantify the effect, and wider impact of intrapartum compromise, as well as the underlying mechanisms for it. After a poor outcome related to intrapartum care parents and healthcare practitioners often strive to understand whether the event could have been predicted and/or prevented. This can be difficult to answer, at least partly related to the heterogeneous fetal response to perinatal asphyxia. Mothers and the maternity service are increasingly encouraged to personalize care and their choices around the birth process, however the information required to guide these choices is most often missing. This makes it difficult for women and professionals to make an informed choice about their care, including the safest mode of birth for them and their baby.

Aim of the study: Identifying antenatal and intrapartum risk factors associated with neonatal hypoxic ischemic encephalopathy.

DETAILED DESCRIPTION:
Antenatal, perinatal and postpartum data will be documented from the medical notes and from parental reports including;

* Booking factors (maternal age, smoking, parity, previous lower segment caesarean section (LSCS), multiple births)
* Antenatal factors (preeclampsia, gestational diabetes, prelabor abruption, placenta previa, oligohydramnios, polyhydramnios, threatened preterm labor, gender, concerns of IUGR infant)
* Labor factors (induction of labor, pre-labor rupture of membranes, planned LSCS, gestation at birth, presentation, prelabor breech, breech delivery, duration of ruptured membranes).
* Infant characteristics included GA, gender, birth weight (BW), head circumference, and multiplicity.
* Clinical signs, examination findings and laboratory data also will be included. Most covariates will be extracted from patient's notes, routine data collection or as part of a routine clinical database.

Data will be processed and analyzed using SPSS software and the results will be processed in tables and figures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of neonatal encephalopathy(e.g. irritability, decreased responsiveness, coma, seizures, hypotonia, abnormal primitive reflexes, apnea, feeding disturbance, and abnormal cry), NICU admission, full-term infant with poor condition at birth (5-minute Apgar score <7) and/or need for major resuscitation.

Exclusion Criteria:

* Preterm infant, full term infants with birth asphyxia but with congenital malformations or chromosomal abnormalities, infant of diabetic mother and CNS infections are excluded from the study.

Ages: 24 Hours to 28 Days | Sex: All
Age Groups: Child
Study Population: Full term infants with clinic linical signs of neonatal encephalopathy(e.g. irritability, decreased responsiveness, coma, seizures, hypotonia, abnormal primitive reflexes, apnea, feeding disturbance, and abnormal cry), NICU admission, full-term infant with poor condition at birth (5-minute Apgar score <7) and/or need for major resuscitation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Antenatal and intrapartum risk factors associated with neonatal hypoxic ischemic encephalopathy. | Baseline
  Antenatal, perinatal and postpartum data will be documented from the medical notes and from parental reports including;
  * Booking factors (maternal age, smoking, parity, previous lower segment caesarean section (LSCS), multiple births)
  * Antenatal factors (preeclampsia, gestational diabetes, prelabor abruption, placenta previa, oligohydramnios, polyhydramnios, threatened preterm labor, gender, concerns of IUGR infant)
  * Labor factors (induction of labor, pre-labor rupture of membranes, planned LSCS, gestation at birth, presentation, prelabor breech, breech delivery, duration of ruptured membranes).
  * Infant characteristics included GA, gender, birth weight (BW), head circumference, and multiplicity.
  * Clinical signs, examination findings and laboratory data also will be included. Most covariates will be extracted from patient's notes, routine data collection or as part of a routine clinical database.

REFERENCES:
- [Background] Glass HC. Hypoxic-Ischemic Encephalopathy and Other Neonatal Encephalopathies. Continuum (Minneap Minn). 2018 Feb;24(1, Child Neurology):57-71. doi: 10.1212/CON.0000000000000557. PMID 29432237
- [Background] Simiyu IN, Mchaile DN, Katsongeri K, Philemon RN, Msuya SE. Prevalence, severity and early outcomes of hypoxic ischemic encephalopathy among newborns at a tertiary hospital, in northern Tanzania. BMC Pediatr. 2017 May 25;17(1):131. doi: 10.1186/s12887-017-0876-y. PMID 28545428
- [Background] Qureshi AM, ur Rehman A, Siddiqi TS. Hypoxic ischemic encephalopathy in neonates. J Ayub Med Coll Abbottabad. 2010 Oct-Dec;22(4):190-3. PMID 22455295
- [Background] Odd D, Heep A, Luyt K, Draycott T. Hypoxic-ischemic brain injury: Planned delivery before intrapartum events. J Neonatal Perinatal Med. 2017;10(4):347-353. doi: 10.3233/NPM-16152. PMID 29286930